CLINICAL TRIAL: NCT07079397
Title: The Integration Pattern of Non-Animal Stabilized Hyaluronic Acid (NASHA)- and Optimum Balance Technology (OBT)-Based Fillers: An Ultrasound and Magnetic Resonance Imaging (MRI) Study
Brief Title: Hyaluronic Acid Filler Migration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAL-2025-MIG-67
Record Dates: First submitted 2025-05-29; First posted 2025-07-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aesthetic
Keywords: Hyaluronic Acid; Fillers; Facial Assessment; Migraion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Restylane Injectables (Other): All adult participants (>18 years)
  Interventions: Device: Restylane Injectables

INTERVENTIONS:
Device: Restylane Injectables — Participants will receive pan-facial treatment in at least one facial area using a Restylane NASHA product and at least one different facial area using Restylane OBT product. Participants will undergo three (3) scheduled MRI scans thoughout the duration of the study post HA injections.

SUMMARY:
Soft tissue filler injections continue to grow in popularity as a method of facial rejuvenation, including volume restoration and contour enhancement.

Many different hyaluronic acid (HA)-based fillers are available on the market and differ in terms of their physical and chemical properties, which results in families of fillers (e.g., Non-Animal Stabilized Hyaluronic Acid - NASHA vs. Optimal Balance Technology - OBT) with different tissue integration patterns. It has been proposed that the properties of fillers significantly influences their tendency to migrate. More specifically, thick fillers may be less prone to migration compared to fluid fillers. However, a detailed knowledge of facial anatomy, safer injection techniques, and careful product selection based on filler qualities may be preventive measures for filler migration.

The goal of this study is to describe the short and intermediate-term product distribution/integration patterns of NASHA and OBT-based fillers, and to evaluate the evidence (if any) of filler migration from the intended site of injection.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, male or female participants 18 years of age and older;
2. Participants with established facial volume loss and/or contour deficits;
3. Accepted the obligation not to receive any other facial procedures throughout the study duration;
4. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits;
5. No previous facial fillers for 18 months prior to this study;
6. Capable of providing informed consent, approved by an independent ethics committee, prior to the initiation of any screening or study-specific procedures;
7. Participants must be willing and able to comply with procedures required in the protocol.
8. Participants must be in good health as per investigator's judgment based on medical. history.
9. Female participants of childbearing potential must be willing practice at least 1 protocol-specified method of birth control that is effective from Baseline through at least 30 days after the last dose or until the end of study, whichever is longer. Female participants of non-childbearing potential do not need to use birth control

Exclusion Criteria:

1. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)];
2. Hypersensitivity to Restylane products, HA filler or amide local anesthetics;
3. Participants presenting with porphyria or any other liver diseases;
4. Inability to comply with follow-up and abstain from facial injections during the study period;
5. Heavy smokers, classified as smoking more than 12 cigarettes per day;
6. History of severe or multiple allergies manifested by anaphylaxis, since drug allergies might preclude optimal management of complications;
7. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
8. Previous facial surgery, including liposuction;
9. Lifetime history of permanent implants in the treatment region;
10. History in the last 18 months of semi-permanent dermal fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation in the treatment region;
11. History or presence of any disease or lesion near or at the treatment area, including inflammation, active or chronic infection, including in the mouth, dentals, head and neck region;
12. Participant has an uncontrolled systemic diseases
13. Participants present with or have a history of any medical condition that may place the participant at increased risk following exposure to hyaluronic acid or interfere with the study evaluation, including:

    * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
    * History of facial nerve palsy
    * Infection or dermatological condition at the treatment injection sites
    * Marked facial dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or excessively photodamaged skin
14. Facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes zoster or any other facial condition that may increase the risk of cutaneous penetration of infective agents;
15. Scars, deformities, piercing, or tattoos in the treatment areas;
16. Facial cancer or precancer (e.g., actinic keratosis);
17. History of radiation therapy to the treatment area;
18. History of bleeding disorders, or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g., Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment;
19. Participants with active immune disorders such as systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, and Hashimoto's thyroiditis, or participants using immunosuppressants;
20. Participants with a tendency to form hypertrophic or keloid scars, or any other healing disorders;
21. Participants with known hypersensitivity to lidocaine or agents structurally related to amide type local anaesthetics (e.g., certain anti-arrhythmics);
22. Participants administered dental block or topical administration of lidocaine within 2 weeks of treatment;
23. Participants with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction;
24. Current remote infections (e.g., urinary tract, sinuses, intestinal tract, oral cavity);
25. Planned dental procedures during the 2-week period before and after filler treatments, including teeth cleaning, tooth extraction and gum grafts.
26. Planned COVID-19 vaccinations during the 2-week period before and after filler treatments.
27. History of cystic acne (for those that will be treated in the chin region).
28. Female participants that is pregnant or breastfeeding and is considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study medical device or until the end of study, whichever is longer
29. Anticipated need for surgery or hospitalization during the course of the study
30. History of other treatment/procedure that, in the treating investigator's opinion, would interfere with the study injections and/or study assessments or exposes the participant to undue risk by study participation.
31. Contraindications for Magnetic Resonance Imaging (MRI) such as:

    * Implanted pacemakers or defibrillators
    * Metallic implants of any kind including cochlear implants and orthodontics
    * Claustrophobia
    * Pregnancy
    * Loud noises

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate evidence (if any) of filler migration from the intended site of injection for NASHA and OBT-based fillers, as visualized by high resolution MRI. | Baseline (post optimal correction), Week 12 and Week 24
  High resolution MRI will determine presence of filler migration. Migration will be assessed radiologically and defined as the presence of identifiable product in anatomical regions outside the treatment area (where the product was initially placed) using a dichotomous qualitative response "yes/no".

SECONDARY OUTCOMES:
Number of particpants assessed as having proudct distribution past the area of injection. Assesment will be determined clincially by a qualified physician. | Baseline (post optimal correction), Week 12 and Week 24
  Physician evaluation will determine the distribution/integration patterns of NASHA and OBT-based fillers through palpable assessment in whcih the physician will use a binary "yes" or "no" responde to denote filler migration from the area of original placemement.
Number of particpants assessed as having proudct distribution past the area of injection. Assesment will be made uisng ultrasoundimaging | Baseline (post optimal correction), Week 12 and Week 24
  Ultrasound evaluation will determine the distribution/integration patterns of NASHA and OBT-based fillers through visual changes to position of filler deposition.

OTHER OUTCOMES:
Evaluate the frequncy of advese events (safety) of pan-facial HA injections. | Baseline to Week 24
  Adverse events (safety) realted to pan-facial injections using NASHA and OBT based products will be determined by the frequency and severity of Adverse Events (AEs):
  1. Physician reported
  2. Participant reported

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevan Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No